CLINICAL TRIAL: NCT00866905
Title: Phase II Study of Ixabepilone and Cyclophosphamide as Neoadjuvant Therapy in HER2-Negative Breast Cancer
Brief Title: Ixabepilone and Cyclophosphamide as Neoadjuvant Therapy in HER-2 Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 133
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Results first posted 2014-11-27 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Ixabepilone; Ixempra; Cyclophosphamide; Cytoxan; Neoadjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ixabepilone/Cyclophosphamide (Experimental): Systemic Therapy followed by surgery and possible radiation therapy
  Interventions: Drug: Ixabepilone; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Ixabepilone — 40 mg/m2 IV infusion over 3 hours on day 1 of a 21 day cycle for 6 cycles
  Other Names: Systemic therapy; Ixempra
Drug: Cyclophosphamide — 600 mg/m2 IV infusion per institutional guidelines on day 1 of a 21 day cycle for 6 cycles
  Other Names: Systemic therapy; Cytoxan

SUMMARY:
We propose to evaluate ixabepilone in combination with cyclophosphamide for the neoadjuvant treatment of locally advanced breast cancer. In this regimen, ixabepilone is substituted for docetaxel, since preclinical and clinical

studies suggest that ixabepilone is more active than either docetaxel or paclitaxel. The combination of ixabepilone and cyclophosphamide could further improve the efficacy of non-anthracycline neoadjuvant therapy.

DETAILED DESCRIPTION:
In this study, patients with early stage, HER2-negative breast cancer will receive neoadjuvant treatment with ixabepilone and cyclophosphamide given every three weeks for a total of six cycles. Following surgery patients with hormone receptor-positive tumors will receive anti-estrogen treatment. Patients may receive local regional radiation therapy after surgery per institutional guidelines at the investigator's discretion. Baseline tumor tissue and tumor tissue removed at the time of surgery will be tested by Oncotype Detailed Description (DX) assay to determine whether it is predictive of response to this neoadjuvant treatment regimen. This study will be one of the first investigations of the combination of ixabepilone and cyclophosphamide as neoadjuvant treatment for HER2-negative breast cancer. It will examine this treatment regimen for potential advantages gained from substitution of ixabepilone for a taxane and use of non-anthracycline agents.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, age ≥18 years.
2. Histologically confirmed invasive adenocarcinoma of the breast.
3. Primary palpable disease confined to a breast and axilla on

   physical examination. For patients without clinically suspicious

   axillary adenopathy, the primary tumor must be larger than 2 cm

   in diameter by physical exam or imaging studies (clinical T2-T3,

   N0-N1, M0). For patients with clinically suspicious axillary

   adenopathy, the primary breast tumor can be any size (clinical

   T1-3, N1-2, M0). (T1N0M0 lesions are excluded.)
4. Patients without clearly defined palpable breast mass or axillary

   lymph nodes but radiographically measurable tumor masses are

   acceptable. Accepted procedures for measuring breast disease

   are mammography, MRI, and breast ultrasound. This will need to

   be re-evaluated after 3 cycles and prior to surgery.
5. Eastern Cooperative Oncology Group performance status (ECOG

   PS) 0-2.
6. No metastatic disease, as documented by complete staging workup

   * 6 weeks prior to initiation of study treatment.
7. No previous treatment for breast cancer.
8. HER2-negative tumor status. HER2-negative is defined as:

   * Immunohistochemical (IHC) 0, IHC 1+ OR
   * IHC 2+ or IHC 3+ must be confirmed as FISH (fluorescence in situ

   hybridization) negative (defined by ratio <2.2).
9. Adequate hematologic function with:

   * Absolute neutrophil count (ANC) >1500/μL.
   * Platelets ≥100,000/μL.
   * Hemoglobin ≥10 g/dL.
10. Adequate hepatic function with:

    * Serum bilirubin ≤ the institutional upper limit of normal (ULN).
    * Aspartate aminotransferase (AST) ≤2.5 x institutional ULN.
    * Alanine aminotransferase (ALT) ≤2.5 x institutional ULN.
11. Adequate renal function with serum creatinine ≤1.5 x ULN.
12. Estrogen and progesterone receptor status in the primary tumor

    known or pending at the time of study registration.
13. Knowledge of the investigational nature of the study and ability to

    provide consent for study participation.
14. For patients who had, or will have sentinel lymph node and/or

    axillary dissection prior to initiation of study treatment, completion

    at least 4 weeks prior to starting study treatment and well-healed

    wound
15. Bilateral, synchronous breast cancer is allowed if one primary

    tumor meets the inclusion criteria.
16. Sufficient archived breast tumor specimen available at baseline

for the Oncotype DX assay.

-

Exclusion Criteria:

1. Inflammatory breast cancer.
2. Peripheral neuropathy (motor or sensory) ≥ grade 1 by the

   Common Terminology Criteria for Adverse Events version 3.0

   (CTCAE v 3.0).
3. Prior radiation that included ≥30% of major bone marrow containing

   areas (pelvis, lumbar, spine).
4. Chronic use of cytochrome P450 (CYP) 3A4 inhibitors and use of

   the following strong CYP3A4 inhibitors: ketoconazole,

   itraconazole, clarithromycin, atazanavir, nefazodone, saquinavir,

   telithromycin, ritonavir, amprenavir, indinavir, nelfinavir,

   delavirdine, and voriconazole. Use of these agents should be

   discontinued at least 72 hours prior to initiation of study treatment.
5. Chemotherapy within 5 years of starting study treatment except

   for low doses of agents used for anti-inflammatory indications

   such as rheumatoid arthritis, psoriasis, and connective tissue

   disorders. Although such doses and schedules cannot result in

   myelosuppression, patients must discontinue this therapy while

   they are receiving study treatment.
6. Known or suspected hypersensitivity to Cremophor®EL

   (polyoxyethylated castor oil) or a drug formulated in

   Cremophor®EL such as paclitaxel, or any other agent given in the

   course of this study.
7. Pregnancy or breast-feeding. A negative serum pregnancy test

   within 7 days prior to first study treatment (Day 1, Cycle 1) for all

   women of childbearing potential is required. Patients of

   childbearing potential must agree to use a birth control method

   that is approved by their study physician while receiving study

   treatment and for 3 weeks after their last dose of study treatment.

   Patients must agree to not breast-feed while receiving study

   treatment.
8. Concurrent treatment with an ovarian hormonal replacement

   therapy or with hormonal agents such as raloxifene, tamoxifen or

   other selective estrogen receptor modulator (SERM). Patients

   must have discontinued use of such agents prior to beginning

   study treatment.
9. History of malignancy treated with curative intent within the

   previous 5 years with the exception of skin cancer, cervical

   carcinoma in situ, or follicular thyroid cancer. Patients with

   previous invasive cancers (including breast cancer) are eligible if

   the treatment was completed more than 5 years prior to initiating

   current study treatment, and there is no evidence of recurrent

   disease.
10. Uncontrolled intercurrent illness including (but not limited to)

    ongoing or active infection.
11. Chronic treatment with corticosteroid unless treatment was begun

    >6 months prior to study treatment and is at a low dose (≤20 mg

    methylprednisolone or equivalent).
12. Use of any investigational agent within 30 days of administration

    of the first dose of study drug.
13. Requirement for radiation therapy concurrent with neoadjuvant

    study chemotherapy.
14. Concurrent treatment with any anti-cancer therapy other than

    those agents used in this study.
15. Inability or unwillingness to comply with study procedures

    including follow-up visits.
16. Mental condition or psychiatric disorder that would prevent patient

    comprehension of the nature, scope, and possible consequences

    of the study or that would limit compliance with study

    requirements.
17. Any other disease(s), metabolic dysfunction, or findings from a

physical examination or clinical laboratory test result that would

cause reasonable suspicion of a disease or condition that

contraindicates the use of study drugs, that may affect the

interpretation of the results, or that renders the patient at high risk

from treatment complications

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-04; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A Yardley, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (20):
- United States (20):
  - Aventura Medical Center, Aventura, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Providence Medical Group, Terre Haute, Indiana
  - Mercy Hospital, Portland, Maine
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Methodist Cancer Center, Omaha, Nebraska
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Family Cancer Center, Collierville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Virginia Cancer Institute, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixabepilone/Cyclophosphamide: Ixabepilone: 40 mg/m2 via intraveous (IV) infusion over 3 hours
  Cyclophosphamide: 600 mg/m2 via IV infusion per institutional guidelines
Period: Overall Study
Arm/Group | Ixabepilone/Cyclophosphamide
Started | 168
Completed | 135
Not Completed | 33

BASELINE CHARACTERISTICS:
Groups:
- Arm/Group 1: All patients who received at least one dose of treatment.
Arm/Group | Arm/Group 1
Number analyzed (Participants) | 168
Age, Continuous [Median (Full Range); unit: Years] | 53 [30 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 168

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate (pCR)
Description: Pathologic complete response (pCR) rate will be determined by the pathologic evaluation of breast and lymph node samples collected at the time of surgery. pCR is defined as no residual disease in breast or lymph nodes in resected tissue samples.
Time Frame: 6 months
Population: To be evaluable, patients had to undergo surgery after neoadjuvant therapy. Out of 168 patients, only 161 patients underwent surgery after neoadjuvant therapy and were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Ixabepilone/Cyclophosphamide
Number analyzed (Participants) | 161
participants | 27

2. Secondary Outcome: Absence of Grade-4 Non-hematologic Toxicity Excluding, Alopecia, Nausea, Vomiting and Bone Pain
Description: Non hematologic treatment-related grade 4 toxicities measured according to CTCAE 3.0
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Ixabepilone/Cyclophosphamide
Number analyzed (Participants) | 168
participants
  Fatigue | 1
  Peripheral neuropathy | 1
  Arthralgia/myalgia | 1

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) determined as the time between day 1 cycle 1 to the date of death from any cause. The percentage of patients who were alive at 3 years, estimated by Kaplan Meier method as the probability of being event free at 3 years is reported here.
Time Frame: 36 months
Population: All patients who received a dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Ixabepilone/Cyclophosphamide
Number analyzed (Participants) | 168
percentage of participants | 90

4. Secondary Outcome: Disease Free Survival
Description: Defined as the time between Day 1 Cycle 1, and date of first documented recurrence, initiation of additional chemotherapy, or death.
Time Frame: 36 Months
Population: All patients who received a dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone/Cyclophosphamide
Number analyzed (Participants) | 168
months | NA [NA to NA] — Median and 95% confidence interval were not estimable by Kaplan-Meier method due to insufficient observed events.

ADVERSE EVENTS:
Groups:
- Ixabepilone/Cyclophosphamide: All patients who received a dose of study treatment
Arm/Group | Ixabepilone/Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 6/168
Other Adverse Events (participants affected / at risk) | 167/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone/Cyclophosphamide (N=168)
DEPRESSION (Psychiatric disorders) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3)
PERIPHERAL NEUROPATHY (Nervous system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone/Cyclophosphamide (N=168)
ABDOMINAL PAIN (Gastrointestinal disorders) | 14 (29)
ALLERGIC REACTION (Immune system disorders) | 10 (10)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 15 (38)
ALOPECIA (Skin and subcutaneous tissue disorders) | 100 (390)
ANEMIA (Blood and lymphatic system disorders) | 118 (430)
ANOREXIA (Metabolism and nutrition disorders) | 41 (92)
ANXIETY (Psychiatric disorders) | 25 (79)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 87 (290)
ASTHENIA (Musculoskeletal and connective tissue disorders) | 17 (30)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 18 (34)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 16 (26)
BREAST PAIN (Reproductive system and breast disorders) | 15 (34)
CHEST PAIN (General disorders) | 9 (16)
CONSTIPATION (Gastrointestinal disorders) | 60 (175)
COUGH (Respiratory, thoracic and mediastinal disorders) | 35 (58)
DEHYDRATION (Metabolism and nutrition disorders) | 10 (12)
DEPRESSION (Psychiatric disorders) | 17 (40)
DIARRHEA (Gastrointestinal disorders) | 60 (127)
DIZZINESS (Nervous system disorders) | 23 (41)
DYSPEPSIA (Gastrointestinal disorders) | 32 (88)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 26 (39)
EDEMA (General disorders) | 14 (32)
FATIGUE (General disorders) | 136 (547)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 12 (15)
FEVER (General disorders) | 16 (18)
HEADACHE (Nervous system disorders) | 38 (95)
HOT FLASHES (Vascular disorders) | 30 (79)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 14 (31)
HYPERTENSION (Vascular disorders) | 13 (28)
INFECTION (Infections and infestations) | 13 (18)
INSOMNIA (Psychiatric disorders) | 48 (145)
LEUKOPENIA (Blood and lymphatic system disorders) | 128 (457)
MUCOSITIS (Gastrointestinal disorders) | 17 (31)
MYALGIA (Musculoskeletal and connective tissue disorders) | 55 (168)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 12 (27)
NAUSEA (Gastrointestinal disorders) | 102 (297)
NEUTROPENIA (Blood and lymphatic system disorders) | 127 (457)
PAIN (General disorders) | 13 (23)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 40 (96)
PARESTHESIA (Nervous system disorders) | 13 (34)
PERIPHERAL NEUROPATHY (Nervous system disorders) | 117 (399)
PRURITUS (Skin and subcutaneous tissue disorders) | 11 (22)
Pain (General disorders) | 21 (37)
RASH (Skin and subcutaneous tissue disorders) | 29 (53)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 10 (11)
TASTE ALTERATION (Nervous system disorders) | 35 (122)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 56 (136)
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 11 (16)
VOMITING (Gastrointestinal disorders) | 32 (54)
WEIGHT LOSS (Investigations) | 11 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from the date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish results until 18 mos. after the trial has been completed at all sites.